CLINICAL TRIAL: NCT05845788
Title: Comparison of the Intraoperative and Postoperative Effects of Ultrasound-guided Erector Spina Plane Block and Posterior Quadratus Lumborum Block in Patients Undergoing Lumbar Stabilization Surgery
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Nihal Gökbulut Özaslan, Principal Investigator, Ankara City Hospital Bilkent
Other Study IDs: E1-23-.3166
Record Dates: First submitted 2023-03-09; First posted 2023-05-06 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Postprocedural Analgesia; Opioid Consumption; Erector Spina Plan Block; Quadratus Lumborum Block

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Erector Spina Plan Block Group (Group E): Patients who underwent erector spina plane block before initiation of surgery after induction of anesthesia
  Interventions: Procedure: Peripheral nerve block
- Posterior Quadratus Lumborum Block Group ( Group Q): Patients who underwent posterior quadratus lumborum block block before initiation of surgery after induction of anesthesia
  Interventions: Procedure: Peripheral nerve block

INTERVENTIONS:
Procedure: Peripheral nerve block — Ultrasound guided peripheral nerve block

SUMMARY:
The investigators aimed to compare the effects of ultrasound guided erector spina plan block and posterior quadratus lumborum block on intraoperative and postoperative opioid consumption in patients who will undergo short segment lumbar stabilization surgery.

DETAILED DESCRIPTION:
All participants will be monitored with ECG, SpO2, non-invasive blood pressure. In induction, 1mg/kg 2% lidocaine, 2-3mg/kg propofol, 1mcg/kg fentanyl, 2mg midazolam, 0.6 mg/kg rocuronium will be used. Anesthesia depth will be monitored with BIS (bispectral index), and anesthesia will be maintained with 50% oxygen-air mixture and sevoflurane. After patient intubation, invasive artery cannulation will be performed on the non-dominant hand, and the patients will be placed in a prone position. 20 cc bupivacaine of 0.25% will be administered to both regions bilaterally, by following the rules of asepsis, with a 10 cm pajunk needle accompanied by USG, the needle site will be confirmed with 3 mm saline.

BIS will be kept in the range of 40-50 throughout the case, and invasive arterial monitoring will be performed. 1 g paracetamol, 1 mg/kg tramadol and 4 mg ondansetron will be administered to the patients 30 minutes before the end of the surgery.

After appropriate extubation and wakefulness, patients will be transferred to the postoperative anesthesia care unit (PACU), where they will be followed for 24 hours.

An intravenous (IV) patient-controlled analgesia device (PCA) containing 100ml of tramadol at a concentration of 4mg/cc will be inserted. No infusion will be given, and the bolus dose will be set to 20mg, with a lock time of 20 minutes. In the postoperative period, 50 mg of dexketoprofen will be administered every 8 hours.

VAS values, vital signs, and possible opioid side effects of the patients at 0, 1, 2, 6, 12 and 24 hours will be recorded. After completing 24 hours, the patient will be separated from the IV PCA device and transferred to the service.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo lumbar stabilization operation
* Between the ages of 18-65
* Both genders
* ASA I-III risk group

Exclusion Criteria:

* Patients who did not accept the study
* Patients younger than 18 years old
* Patients older than 65 years
* Patients with an ASA score greater than III
* Patients with an active infection in the area to be blocked
* Patients with a long bleeding time
* Those who are pregnant
* Patients with kidney failure
* Patients with liver failure
* Patients with BMI<18 and BMI>30
* Those who are allergic to local anesthetics
* Patients who have had previous lumbar surgery
* Uncooperative or mentally retarded patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will undergo lumbar stabilization operation under general anesthesia in Ankara Bilkent City Hospital Operating Room, between the ages of 18-65, both genders, and in the ASA I-III risk group will be included in the study.
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-08-02 (Actual); Study Completion 2023-08-02 (Actual)

PRIMARY OUTCOMES:
İntraoperative remifentanil consumption | At the end of the intraoperative period
  The investigators aimed to compare intraoperative remifentanil consumption of two groups
Postoperative tramadol consumption | The investigators will record at postoperative 0. hour
  The investigators aimed to compare postoperative tramadol consumption of two groups
Postoperative tramadol consumption | The investigators will record at postoperative 1. hour
  The investigators aimed to compare postoperative tramadol consumption of two groups
Postoperative tramadol consumption | The investigators will record at postoperative 2. hour
  The investigators aimed to compare postoperative tramadol consumption of two groups
Postoperative tramadol consumption | The investigators will record at postoperative 6. hour
  The investigators aimed to compare postoperative tramadol consumption of two groups
Postoperative tramadol consumption | The investigators will record at postoperative 12. hour
  The investigators aimed to compare postoperative tramadol consumption of two groups
Postoperative tramadol consumption | The investigators will record at postoperative 24. hour
  The investigators aimed to compare postoperative tramadol consumption of two groups

SECONDARY OUTCOMES:
Postoperative nausea and vomiting | The investigators will record within 24 hours postoperatively.
  Whether there is postoperative nausea and vomiting will be questioned by the investigators. Yes or no will be marked in the table.
Postoperative pruritus | The investigators will record within 24 hours postoperatively.
  Whether there is postoperative pruritus will be questioned by the investigators. Yes or no will be marked in the table.
Postoperative visual analog scale | The investigators will record at postoperative 0. hour
  The investigators aimed to compare patient's visual analog scales of two groups. The visual pain scale is measured with a ruler from 0 to 10 cm. 0 indicates no pain, 10 indicates severe pain.
Postoperative visual analog scale | We will record at postoperative 1. hour
  The investigators aimed to compare patient's visual analog scales of two groups. The visual pain scale is measured with a ruler from 0 to 10 cm. 0 indicates no pain, 10 indicates severe pain.
Postoperative visual analog scale | The investigators will record at postoperative 2. hour
  The investigators aimed to compare patient's visual analog scales of two groups. The visual pain scale is measured with a ruler from 0 to 10 cm. 0 indicates no pain, 10 indicates severe pain.
Postoperative visual analog scale | The investigators will record at postoperative 6. hour
  The investigators aimed to compare patient's visual analog scales of two groups. The visual pain scale is measured with a ruler from 0 to 10 cm. 0 indicates no pain, 10 indicates severe pain.
Postoperative visual analog scale | The investigators will record at postoperative 12. hour
  The investigators aimed to compare patient's visual analog scales of two groups. The visual pain scale is measured with a ruler from 0 to 10 cm. 0 indicates no pain, 10 indicates severe pain.
Postoperative visual analog scale | The investigators will record at postoperative 24. hour
  The investigators aimed to compare patient's visual analog scales of two groups. The visual pain scale is measured with a ruler from 0 to 10 cm. 0 indicates no pain, 10 indicates severe pain.

OTHER OUTCOMES:
Postoperative pulse rate | The investigators will record at postoperative 0. hour
  The investigators aimed to compare patient's pulse rates of two groups.
Postoperative pulse rate | The investigators will record at postoperative 1. hour
  The investigators aimed to compare patient's pulse rates of two groups.
Postoperative pulse rate | The investigators will record at postoperative 2. hour
  The investigators aimed to compare patient's pulse rates of two groups.
Postoperative pulse rate | The investigators will record at postoperative 6. hour
  The investigators aimed to compare patient's pulse rates of two groups.
Postoperative pulse rate | The investigators will record at postoperative 12. hour
  The investigators aimed to compare patient's pulse rates of two groups.
Postoperative pulse rate | The investigators will record at postoperative 24. hour
  The investigators aimed to compare patient's pulse rates of two groups.
Postoperative oxygen saturation | The investigators will record at postoperative 0. hour
  The investigators aimed to compare patient's intraoperative oxygen saturations of two groups
Postoperative oxygen saturation | The investigators will record at postoperative 1. hour
  The investigators aimed to compare patient's intraoperative oxygen saturations of two groups
Postoperative oxygen saturation | The investigators will record at postoperative 2. hour
  The investigators aimed to compare patient's intraoperative oxygen saturations of two groups
Postoperative oxygen saturation | The investigators will record at postoperative 6. hour
  The investigators aimed to compare patient's intraoperative oxygen saturations of two groups
Postoperative oxygen saturation | The investigators will record at postoperative 12. hour
  The investigators aimed to compare patient's intraoperative oxygen saturations of two groups
Postoperative oxygen saturation | The investigators will record at postoperative 24. hour
  The investigators aimed to compare patient's intraoperative oxygen saturations of two groups
Postoperative sistolic and diastolic blood pressure | The investigators will record at postoperative 0. hour
  The investigators aimed to compare patient's blood pressures of two groups
Postoperative sistolic and diastolic blood pressure | The investigators will record at postoperative 1. hour
  The investigators aimed to compare patient's blood pressures of two groups
Postoperative sistolic and diastolic blood pressure | The investigators will record at postoperative 2. hour
  The investigators aimed to compare patient's blood pressures of two groups
Postoperative sistolic and diastolic blood pressure | The investigators will record at postoperative 6. hour
  The investigators aimed to compare patient's blood pressures of two groups
Postoperative sistolic and diastolic blood pressure | The investigators will record at postoperative 12. hour
  The investigators aimed to compare patient's blood pressures of two groups
Postoperative sistolic and diastolic blood pressure | The investigators will record at postoperative 24. hour
  The investigators aimed to compare patient's blood pressures of two groups.
Change from baseline systolic and diastolic blood pressure | The investigators will record every 10 minutes until the end of the surgery
  The investigators aimed to compare patient's blood pressures change of two groups
Change from baseline pulse rate | The investigators will record every 10 minutes until the end of the surgery
  The investigators aimed to compare patient's intraoperative pulse rates change of two groups
Change from baseline oxygen saturation | The investigators will record every 10 minutes until the end of the surgery
  The investigators aimed to compare patient's baseline oxygen saturation change of two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital, Bilkent, Ankara, Cankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Qiu Y, Zhang TJ, Hua Z. Erector Spinae Plane Block for Lumbar Spinal Surgery: A Systematic Review. J Pain Res. 2020 Jul 1;13:1611-1619. doi: 10.2147/JPR.S256205. eCollection 2020. PMID 32669870
- [Background] Dhanjal ST, Tonder S. Quadratus Lumborum Block. 2023 Aug 14. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK537212/ PMID 30725897
- [Background] Elsharkawy H, El-Boghdadly K, Barrington M. Quadratus Lumborum Block: Anatomical Concepts, Mechanisms, and Techniques. Anesthesiology. 2019 Feb;130(2):322-335. doi: 10.1097/ALN.0000000000002524. No abstract available. PMID 30688787
- [Background] Kang R, Lee S, Kim GS, Jeong JS, Gwak MS, Kim JM, Choi GS, Cho YJ, Ko JS. Comparison of Analgesic Efficacy of Erector Spinae Plane Block and Posterior Quadratus Lumborum Block in Laparoscopic Liver Resection: A Randomized Controlled Trial. J Pain Res. 2021 Dec 11;14:3791-3800. doi: 10.2147/JPR.S343366. eCollection 2021. PMID 34924770